

# PROTOCOL A4061079

A PHASE 1B, OPEN LABEL, DOSE FINDING STUDY TO EVALUATE SAFETY, PHARMACOKINETICS AND PHARMACODYNAMICS OF AXITINIB (AG-013736) IN COMBINATION WITH PEMBROLIZUMAB (MK-3475) IN PATIENTS WITH ADVANCED RENAL CELL CANCER

# **Statistical Analysis Plan**

(SAP)

Version: 1.1

**Author:** PPD

**Date:** July 14, 2015

# **TABLE OF CONTENTS**

| 1. AMENDMENTS FROM PREVIOUS VERSION(S) | 4 |
|---|---|
| 2. INTRODUCTION | 4 |
| 2.1. Study Design | 4 |
| 2.2. Study Objectives | 5 |
| 2.2.1. Primary Objective | 5 |
| 2.2.2. Secondary Objectives | 5 |
| 3. INTERIM ANALYSES, FINAL ANALYSES, AND UNBLINDING | 6 |
| 4. HYPOTHESES AND DECISION RULES | 6 |
| 4.1. Statistical Hypotheses | 6 |
| 4.2. Statistical Decision Rules | 6 |
| 5. ANALYSIS POPULATIONS | 6 |
| 5.1. Safety Analysis Set | 6 |
| 5.2. Per Protocol Analysis Set (Evaluable for DLT) | 7 |
| 5.3. Response Evaluable Analysis Set | 7 |
| 5.4. PK Analysis Set | 7 |
| 5.5. Biomarker Analysis Set | 7 |
| 5.6. Treatment Misallocations | 7 |
| 5.7. Protocol Deviations | 7 |
| 6. ENDPOINTS AND COVARIATES | 8 |
| 6.1. Efficacy Endpoints | 8 |
| 6.2. Safety Endpoints | 9 |
| 6.2.1. Dose Limiting Toxicity (DLT) (Primary Endpoint for Dose Finding Cohorts) | 9 |
| 6.2.2. Adverse Events | 10 |
| 6.2.3. Laboratory Abnormalities | 10 |
| 6.3. PK Endpoints | 10 |
| 6.4. Biomarker Endpoints | 11 |
| 6.5. Covariates | 11 |
| 7. HANDLING OF MISSING VALUES | 11 |
| 7.1. Missing Dates | 11 |
| 7.2. Missing Efficacy Endpoint Values | 11 |
| 7.3 Pharmacokinetics | 11 |

| 7.4. Pharmacodynamic Biomarkers | 13 |
|---|---|
| 8. STATISTICAL METHODOLOGY AND STATISTICAL ANALYSES | 13 |
| 8.1. Statistical Methods | 13 |
| 8.1.1. Statistical Methods for Dose Escalation: Up-and-Down Matrix Design with the mTPI Method | 13 |
| 8.1.2. Methods for Estimating the MTD | 14 |
| 8.1.3. Sample Size Determination | 14 |
| 8.2. Statistical Methods for Different Types of Endpoints | 15 |
| 8.3. Statistical Analyses | 15 |
| 8.3.1. Standard Analyses | 15 |
| 8.3.2. Analysis of Efficacy Endpoints | 16 |
| 16 | |
| 8.3.3. Analysis of Safety Endpoints | 16 |
| 8.3.3.1. Analysis of Primary Endpoint | 17 |
| 8.3.3.2. Analysis of Secondary Safety Endpoint | 17 |
| 8.3.4. Analysis of Pharmacokinetics | 20 |
| 8.3.4.1. Pharmacokinetic Analysis of MK-3475 and Axitinib | 21 |
| 8.3.4.2. Effect of MK-3475 on Axitinib Pharmacokinetics | 22 |
| 8.3.4.3. Immunogenecity Assessment | 22 |
| 8.3.4.4. Population Pharmacokinetic Analysis or PK/PD Modeling . | 22 |
| 8.3.5. Analysis of Biomarker Endpoints | 22 |
| 8.4. Summary of Secondary Efficacy Analyses | 24 |
| 9. REFERENCES | 25 |
| 10. APPENDICES | 26 |
| Appendix 1. Programming Specifications for AE Analyses | 26 |
| Appendix 2. Study Specific Information for Efficacy | 31 |
| Appendix 3. RECIST 1.1 | 32 |
| Appendix 4 Detailed Dose Escalation/De-Escalation Scheme | 35 |

# 1. AMENDMENTS FROM PREVIOUS VERSION(S)

- Specifies analyses of safety data (adverse events and laboratory tests) which includes the period from the start of treatment with the axitinib + MK-3475 combination (CD1).
- Clarified language regarding analysis sets for efficacy endpoints. Clarified that data from patients treated at the MTD in the dose escalation and dose expansion portions of the study will be pooled for the secondary safety and efficacy analyses.
- Removed supportive efficacy analysis.

#### 2. INTRODUCTION

This document describes the planned statistical analyses for Protocol A4061079. This analysis plan is meant to supplement the study protocol. In this document, any text taken directly from the protocol is *italicized*.

Any deviations from this main analysis plan will be described in the Clinical Study Report.

# 2.1. Study Design

This is a Phase 1b, open-label, multi-center, multiple-dose, safety, pharmacokinetics (PK) and pharmacodynamic study of axitinib in combination with MK-3475 in adult patients with previously untreated advanced renal cell carcinoma (aRCC). This clinical study will be composed of a Dose Finding Phase and a Dose Expansion Phase. The Dose Finding Phase will estimate the maximum tolerated dose (MTD) in patients with aRCC with clear cell histology who did not receive prior systemic therapy for the advanced disease, using the modified toxicity probability interval (mTPI) method.

The Dose Finding Phase will lead to the identification of an Expansion Test Dose for axitinib in combination with MK-3475 in patients with aRCC who did not receive prior systemic therapy. The Expansion Test Dose will be either the MTD (ie, the highest dose of axitinib and MK-3475 associated with the occurrence of dose limiting toxicities (DLTs) in <33% of patients) or the recommended phase II Dose (RP2D), ie, the highest tested dose that is declared safe and tolerable by the Investigators and Sponsor. Once the Expansion Test Dose is identified, the Dose Expansion Phase will be opened and axitinib in combination with MK-3475 will be tested in patients with previously untreated aRCC.

Anti-tumor activity will be assessed by radiological tumor assessments conducted at baseline, 12 weeks, and every 6 weeks thereafter, using response evaluation criteria in solid tumors (RECIST) version 1.1. In addition, radiological tumor assessments will also be conducted whenever disease progression is suspected (e.g., symptomatic deterioration), and at the time of End of Treatment/Withdrawal (if not done in the previous 6 weeks). Brain CT or MRI scans are required at baseline and when there is a suspected brain metastasis. Bone scan (bone scintigraphy) or <sup>18</sup>F-FDG-PET/CT is required at baseline then every 15 weeks only if bone metastases are present at baseline. Otherwise bone imaging is required only if

new bone metastases are suspected. Bone imaging is also required at the time of confirmation of response for patients who have bone metastases.

MK-3475 and axitinib do not have competing elimination/metabolism pathways, hence an overt PK interaction between the two drugs is not anticipated. However, pharmacokinetic assessments will be conducted in this study to confirm the absence of drug-drug interactions. To understand the PK effects of MK-3475 on axitinib, a 7-day lead-in period with single-agent axitinib will be included prior to Cycle 1 in all patients in the Dose Finding Phase and in at least 8 patients in the Dose Expansion Phases of the study. On the contrary, the administration of single agent MK-3475 to this patient population is not considered in this trial. The effect of axitinib on MK-3475 will be evaluated by comparing MK-3475 trough concentrations at steady-state in the presence of axitinib with those reported for MK-3475 alone in prior studies. MK-3475 has a long half-life (21-28 days) and an increase in trough concentration over time is expected.

Archived tumor biospecimens, and baseline de novo biospecimens from metastatic lesions will be collected for all patients in the dose expansion cohort. Every effort will be made to obtain a second biopsy at the time of first tumor assessment at 12 weeks. Biomarker studies on tumor and blood biospecimens will be carried out to help understand the mechanism of action of the axitinib plus MK-3475 combination, as well as potential mechanisms of resistance. Such results may help in the future development of this combination. Analyses using translational approaches may also result in the identification of potential biomarkers of response to the axitinib plus MK-3475 combination, ultimately leading to the development of a patient selection strategy for further clinical investigation. As such, collection of tumor and blood biospecimens at baseline and on study will be of paramount importance.

# 2.2. Study Objectives

## 2.2.1. Primary Objective

• To assess the safety and tolerability of axitinib in combination with MK-3475 in patients with previously untreated advanced RCC in order to estimate the MTD and select the RP2D.

#### 2.2.2. Secondary Objectives

- To evaluate the overall safety profile of axitinib in combination with MK-3475.
- To assess the anti-tumor activity of axitinib in combination with MK-3475 in patients with advanced RCC in the first-line treatment setting.
- To characterize the PK of axitinib and axitinib plus MK-3475 when administered in combination, and to assess the effect of MK-3475 on the PK of axitinib.
- To characterize, using translational approaches, genes and proteins such as PD-L1, VEGF-A and IL-8 relevant to angiogenisis drug target pathway, renal cell carcinoma biology, and sensitivity/resistance mechanisms to axitinib in combination with MK-3475 in tumor and/or blood.

- To explore the pharmacodynamic effect of axitinib in combination with MK-3475 in blood and tumor by assessment of gene, RNAs and proteins including but not limited to VEGF-A, IL-8 and VEGFR2 and T-cell receptors.
- *To assess the immunogenicity of MK-3475.*

# 3. INTERIM ANALYSES, FINAL ANALYSES, AND UNBLINDING

This is an open label, single-arm trial for which no formal interim analysis is planned. The final analysis of efficacy will be performed approximately 18 months after enrollment of the last subject; however, earlier analyses of the data may be performed for publication and regulatory reporting purposes.

#### 4. HYPOTHESES AND DECISION RULES

## 4.1. Statistical Hypotheses

The emphasis of the final analyses will be on estimation of key summary statistics rather than hypothesis testing.

#### 4.2. Statistical Decision Rules

#### Up-and-Down Matrix Design with the mTPI Method

The dose escalation/de-escalation rules will follow the mTPI method (see Section 8 for a detailed description). Briefly, the mTPI method relies upon a statistical probability algorithm, calculated using data from all patients treated at the same dose level (and not simply those in the current cohort) to determine whether future cohorts should involve dose escalation, no change in dose, or dose de-escalation.

#### Maximum Tolerated Dose Definition

The MTD estimate is the highest dose of axitinib and MK-3475 associated with the occurrence of DLTs in <33% of patients.

#### Dose Expansion Phase Cohorts

Once the MTD (or the RP2D) for the combination has been defined, up to 40 response-evaluable patients with advanced RCC will be enrolled and treated in the Expansion Phase. The expansion phase will confirm the safety and tolerability as well as explore the antitumor activity of axitinib in combination with MK-3475 in patients with previously untreated advanced RCC.

#### 5. ANALYSIS POPULATIONS

#### 5.1. Safety Analysis Set

The safety analysis set includes all enrolled patients who receive at least one dose of axitinib or MK-3475. This is the primary population for all standard analyses.

# 5.2. Per Protocol Analysis Set (Evaluable for DLT)

All enrolled patients who are eligible, receive at least one dose of axitinib and MK-3475, and who either experience DLT during the first two cycles, or complete the observation period for the first two cycles of treatment (6 weeks). Patients who withdraw from study treatment before receiving at least 75% of the planned first two cycles doses of axitinib or two infusions of MK-3475 within the DLT observation period due to reasons other than treatment related adverse events are not evaluable for DLT.

#### 5.3. Response Evaluable Analysis Set

All patients who receive study treatment (at least one dose of axitinib and MK-3475) with an adequate baseline tumor assessment will be considered evaluable for anti-tumor efficacy using standard RECIST 1.1 criteria.

## 5.4. PK Analysis Set

The PK concentration population is defined as all treated patients who have at least 1 concentration of either of the study drugs.

The PK parameter analysis population is defined as all treated patients who have at least 1 of the PK parameters of interest of any of the study drugs.

# 5.5. Biomarker Analysis Set

The biomarker analysis population is defined separately for blood-based and tumor tissue-based biomarkers. The biomarker analysis population includes all enrolled patients who receive at least one dose of any study drug, and have at least one biomarker parameter from the corresponding assay sample with at least one baseline biomarker measurement. The following are the biomarker analysis sets for the purpose of specific PD biomarker analysis:

Serum biomarker analysis set,

Whole blood biomarker analysis set, and

Tumor biomarker analysis set.

#### 5.6. Treatment Misallocations

Not applicable.

#### 5.7. Protocol Deviations

All deviations will be described when they appear and relate to the statistical analyses or analyses populations.

#### 6. ENDPOINTS AND COVARIATES

## 6.1. Efficacy Endpoints

Assessment of response will be made using RECIST version 1.1. All response statuses will be derived from lesion measurement data recorded on the electronic case report forms as provided by the investigator.

Tumor assessments will include all known or suspected disease sites. Imaging may include chest, abdomen and pelvis CT or MRI scans; brain CT or MRI scan for patients with known or suspected brain metastases; bone scan for patients with known or suspected bone metastases.

The same imaging technique used to characterize each identified and reported lesion at baseline will be employed in the following tumor assessments.

Antitumor activity will be assessed through radiological tumor assessments conducted at baseline (screening), at 12 weeks, and every 6 weeks thereafter. In addition, radiological tumor assessments will also be conducted whenever disease progression is suspected (e.g. symptomatic deterioration) and at the time of withdrawal from the treatment (if not done in the previous 6 weeks).

- Objective Response Rate (ORR) is defined as the percent of patients with confirmed complete response (CR) or confirmed partial response (PR) according to the RECIST 1.1, relative to the response evaluable population. Confirmed responses are those that persist on repeat imaging study at least 4 weeks after initial documentation of response. Patients who do not have on-study radiographic tumor re-evaluation or who die, progress, or drop out for any reason prior to reaching a CR or PR will be counted as non-responders in the assessment of ORR. A patient who initially meets the criteria for a PR and then subsequently becomes a confirmed CR will be assigned a best response of CR.
- **Progression Free Survival (PFS)** is defined as the time from the date of first dose of MK-3475 (C1D1) to the date of the first documentation of objective tumor progression or death on-study due to any cause, whichever occurs first. If tumor progression data include more than 1 date, the first date will be used. PFS (in months) will be calculated as (first event date first dose date +1)/30.44.

Patients lacking an evaluation of tumor response after the date of the first dose of MK-3475 (C1D1) will have their event time censored on the date of the first dose unless death occurs prior to 18 weeks (in which case the death is an event).

If patients have at least 1 on-study disease assessment, PFS data will be censored on the date of the last evaluable tumor assessment documenting absence of progressive disease for patients:

Who are alive and progression free at the time of the analysis (note: summaries
will distinguish between subjects still in disease follow-up verses those who have
discontinued);

- Who have documentation of disease progression or death on study after ≥2, consecutive missed tumor assessments (i.e. >18 weeks for the first two assessments and then subsequently >12 weeks after last tumor assessment);
- Who are given anti-tumor treatment other than the study medication prior to documented disease progression or death.

PFS (months) = [progression/death date - date of first dose +1]/30.44

- **Six-month progression-free survival (6m-PFS)** is summarized as a product limit estimator based on the Kaplan-Meier method to account for censored events.
- Twelve-month progression-free survival (12m-PFS) is summarized as a product limit estimator based on the Kaplan-Meier method to account for censored events.
- **Time to Response (TTR)** is defined as the time from first dose of MK-3475 (CID1) to the first documentation of objective tumor response (CR or PR) that is subsequently confirmed. TTR will only be calculated for the subgroup of patients with a confirmed objective tumor response.

TTR (months) = [first date of OR – date of first dose +1]/30.44

• **Duration of Response (DR)** is defined as the time from first documentation of objective tumor response (CR or PR) until the first date that recurrent, progressive disease, or death due to any cause (whichever occurs first) is objectively documented. If tumor progression data include more than 1 date, the first date will be used. Censoring for DR is identical to the censoring rules presented for PFS. DR will only be calculated for the subgroup of patients with a confirmed objective tumor response.

DR (months) = [progression/death date - first date of OR +1]/30.44

• Overall Survival (OS) is defined as the time from the first dose of MK-3475 (C1D1) to the date of death due to any cause. OS will be summarized in the response evaluable population. For patients still alive at the time of the analysis, the OS time will be censored on the last date they were known to be alive. Patients lacking data beyond the day of first dose of study treatment will have their survival times censored at 1 day.

OS (months) = [date of death - date of first dose +1]/30.44

# 6.2. Safety Endpoints

# 6.2.1. Dose Limiting Toxicity (DLT) (Primary Endpoint for Dose Finding Cohorts)

Severity of AEs will be graded according to NCI CTCAE v 4.03. AEs meeting one of the definition criteria in protocol Section 3.1.2 occurring in the DLT observation period (6 weeks post C1D1) which are attributable to one or both study drugs will be classified as DLTs.

#### 6.2.2. Adverse Events

AEs will be characterized by type, frequency, severity (as graded by NCI CTCAE version 4.03), timing, seriousness and relationship to study treatment. Adverse events occurring during the 7 day lead in phase for PK will be summarized separately from adverse events reporting after first dose of MK-3475 (C1D1). Baseline signs and symptoms will be recorded at baseline and then reported as adverse events during the trial if they worsen in severity or increase in frequency.

## **Treatment Emergent Adverse Events**

All deaths and serious AEs, regardless of cause, occurring from start of treatment until 28 days after the last dose will be considered treatment-emergent. All other non-serious AEs occurring after treatment start regardless of cause, will be considered treatment-emergent up until 28 days after the last dose or until start of new anti-cancer treatment, whichever occurs first. Disease progression is not considered a treatment emergent AE unless the patient dies of disease prior to 28 days after the last dose. Events that are continuations of baseline abnormalities are considered treatment emergent AEs only if there is an increase in grade over baseline, or if there is an increase following a decrease during the study.

For subjects with a 7 day lead-in phase for PK, adverse events reported during the lead-in phase will only be considered as treatment emergent for the combination if there is an increase in grade after the first dose of MK-3475 (C1D1) or if there is a decrease and then subsequent increase during treatment with the combination.

#### **Treatment Related Adverse Events**

Treatment emergent AEs with causality related to treatment, as judged by the investigator, will be considered treatment-related. Events that are continuation of baseline abnormalities are not considered treatment- related unless there is an increase in grade, or if there is an increase following a decrease, and the increase is judged by the investigator to be due to treatment

## **6.2.3.** Laboratory Abnormalities

Laboratory abnormalities as characterized by type, frequency, severity (as graded by NCI CTCAE v. 4.03) and timing. Abnormalities occurring during the 7 day lead in phase for PK will be summarized separately from abnormalities occurring after first dose of MK-3475 (C1D1).

For summaries of the lead-in PK phase and the treatment period starting at C1D1, baseline will be defined as the last evaluation within 28 days prior to the first dose of axitinib and MK-3475, respectively. For laboratory summaries of the entire treatment period (including by cycle), baseline will be defined as the last evaluation within 28 days prior to the first dose of either axitinib or MK-3475, whichever occurs first.

# 6.3. PK Endpoints

Axitinib pharmacokinetic analysis will be conducted at Pfizer. The MK-3475 pharmacokinetic analysis will be conducted at Merck and results will be shared with Pfizer.

Pharmacokinetic parameters for axitinib:

•  $C_{max}$ ,  $T_{max}$ ,  $AUC_{0-12}$ , CL/F and  $V_z/F$  as data permit.

# 6.4. Biomarker Endpoints

Translational and pharmacodynamic biomarkers will be assessed separately for blood and tumor biopsy specimens. These will include measurements of DNA, RNA or protein markers known or suspected to be of relevance to the mechanism of action, the development of resistance, or the identification of those patients who might benefit from treatment with axitinib and MK-3475 combination. The assessment will include pre- and post-baseline blood level of circulating biomarkers; Circulating markers that may be analyzed include, but may not be limited to soluble proteins/cytokines such as VEGF-A, VEGFR2, IL8 and T-cell receptor expansion.

Archival tumor biospecimens (all patients) and baseline *de novo* biospecimens from metastatic lesions (expansion cohort) will be assessed. Post-baseline assessment may be performed for expansion cohort. Tumor biopsies assessment will include tumor tissue biomarkers (e,g, drug targets such as PD-L1; and other markers, such as CD68).

#### 6.5. Covariates

None.

## 7. HANDLING OF MISSING VALUES

# 7.1. Missing Dates

In compliance with Pfizer standards, if the day of the month is missing for any date used in a calculation, the 1<sup>st</sup> of the month will be used to replace the missing date unless the calculation results in a negative time duration (e.g., date of resolution cannot be prior to date of onset; if replacing resolution date with the 1<sup>st</sup> of the month results in a negative duration, the resolution date will be set to the onset date.). In this case, the date resulting in 0 time duration will be used. Pfizer standards are also used if both month and day are missing (Jan 1 unless negative time duration). For PFS, TTR, DR and OS, if conventions result in a negative duration, durations will be reset to 1 day.

If the start date is missing for an AE, the AE is considered to be treatment emergent unless the collection date is prior to the treatment start date.

#### 7.2. Missing Efficacy Endpoint Values

For all efficacy analyses no values will be imputed for missing data, except as specified in Section 6.1, where for ORR, patients with no post-baseline tumor evaluations will be counted as non-responders.

#### 7.3. Pharmacokinetics

#### **Concentrations below the limit of quantification:**

In all data presentations (except listings), axitinib concentrations below the limit of quantification (BLQ) will be set to zero. In listings, BLQ values will be reported as "<LLQ", where LLQ will be replaced with the value for the lower limit of quantification for axitinib.

# Deviations, missing concentrations and anomalous values:

For summary tables and plots of median profiles, appropriate summary statistics will be calculated. Concentrations will be set to missing if one of the following cases is true:

- 1. A concentration has been reported as ND (i.e., not done) or NS (i.e., no sample),
- 2. A deviation in sampling time is of sufficient concern or a concentration has been flagged as anomalous by the pharmacokineticist.

Note that summary statistics will not be presented at a particular time point if more than 50% of the data are missing. For analysis of PK concentrations, no values will be imputed for missing data.

## Pharmacokinetic parameters:

Axitinib pharmacokinetic analysis will be conducted at Pfizer. The MK-3475 pharmacokinetic analysis will be conducted at Merck and results will be shared with Pfizer.

Actual PK sampling times (and where possible the actual dosing information) will be used in the derivation of axitinib PK parameters. If a PK parameter cannot be estimated from a subject's concentration data, the parameter will be coded as NC (i.e., not calculated). (Note that NC values will not be generated beyond the day that a subject discontinues).

In summary tables, statistics will be calculated by setting NC values to missing; and statistics will not be presented for a particular treatment if more than 50% of the data are NC. For statistical analyses (i.e., analysis of variance), PK parameters coded as NC will also be set to missing.

If an individual subject has a known biased estimate of a PK parameter (due for example to an unexpected event such as vomiting before allof the drug is absorbed in the body), this will be footnoted in summary tables and will not be included in the calculation of summary statistics or statistical analyses.

For PK analysis, patients will be required to have at least one quantifiable concentration of each drug to be included in the concentration summary. For evaluation of changes in PK of axitinibwhen administered alone vs in combination, only patients with matching pair of PK assessments under both conditions will be included in the PK summary. Patients who have been treated with axitinib for whom drug plasma concentrations (from both PK visits, when administered alone and in combination) are available will be included in average concentration summary.

#### 7.4. Pharmacodynamic Biomarkers

For analysis of pharmacodynamic biomarkers, no values will be imputed for missing data.

Duplicate biomarker (i.e., more than one set of data for a particular visit) is not expected. For continuous data, if duplicate data is received, the results will be averaged and the average value will be used. The average value will be added to the analysis dataset. For non-continuous data, the results will be reviewed by the study team and a representative sample will be selected. The representative sample will be flagged in the analysis dataset.

#### 8. STATISTICAL METHODOLOGY AND STATISTICAL ANALYSES

#### 8.1. Statistical Methods

# **8.1.1. Statistical Methods for Dose Escalation: Up-and-Down Matrix Design with the mTPI Method**

The mTPI design uses a Bayesian statistics framework and a beta/binomial hierarchical model to compute the posterior probability of three dosing intervals that reflect the relative difference between the toxicity rate of each dose level to the target rate (pT = 0.30). If the toxicity rate of the currently used dose level is far smaller than pT, the mTPI will recommend escalating the dose level; if it is close to pT, the mTPI will recommend continuing at the current dose; if it is far greater than pT, the mTPI will recommend de-escalating the dose level. These rules are conceptually similar to those used by the 3+3 design, except the decisions of an mTPI design are based on posterior probabilities calculated under a coherent probability model.

Being a model-based design, mTPI automatically and appropriately tailors dose-escalation and de-escalation decisions for different trials with different toxicity parameters. More importantly, all the dose-escalation decisions for a given trial can be pre-calculated under the mTPI design and presented in a two-way table (Appendix 4). Thus, compared to other advanced model-based designs published in the literature, the mTPI design is logistically less complicated and easier to implement. Recently, a Phase 1 trial based on the mTPI design has been published.<sup>4</sup>

Decision rules are based on calculating unit probability mass (UPM) of three dosing intervals corresponding to under, proper, and over dosing in terms of toxicity. Specifically, the underdosing interval is defined as  $(0; pT-e_1)$ , the over-dosing interval  $(pT+e_2)$ , and the proper-dosing interval  $(pT-e_1, pT+e_2)$ , where  $e_1$  and  $e_2$  are small fractions. Based on the safety profile of axitinib and MK-3475,  $e_1$  is selected as 0.05, and  $e_2$  is selected as 0.03. Therefore, the target dosing interval for the DLT rate is (0.25, 0.33).

The three dosing intervals are associated with three different dose-escalation decisions. The under-dosing interval corresponds to a dose escalation (E), over-dosing corresponds to a dose de-escalation (D), and proper-dosing corresponds to remaining at the current dose (R). Given a dosing interval and a probability distribution, the unit probability mass (UPM) of that dosing interval is defined as the probability of a subject belonging to that dosing interval divided by the length of the dosing interval. The mTPI design calculates the UPMs for the

three dosing intervals, and the one with the largest UPM informs the corresponding dose-finding decision, which is the dose level to be used for future patients. For example, if the under-dosing interval has the largest UPM, the decision will be to escalate, and the next cohort of patients will be treated at the next higher dose level. Ji and collaborators have demonstrated that the decision based on UPM is optimal in that it minimizes a posterior expected loss (ie, minimizes the chance of making a wrong dosing decision)<sup>5</sup>.

The dose-finding component of the trial is completed when at least 10 evaluable patients have been treated at the highest dose with DLT rate < 0.33. It is estimated that approximately 20 DLT evaluable patients have been enrolled to reach10-DLT evaluable patients at the estimated MTD.

# 8.1.2. Methods for Estimating the MTD

The estimated MTD will be the highest tested dose level with a DLT rate <0.33 in 10 DLT evaluable patients. We assume that higher doses of MK-3475 result in higher toxicity rates. But, due to the relatively low number of patients that may be potentially allocated to any dose combination, this assumption may be violated. For example, at the end of the study, the dose combination (MK-3475 2 mg /kg q3wks, axitinib 5 mg BID) may have a higher proportion of observed toxicities than, say, (MK-3475 1 mg /kg q3wks, axitinib 5 mg BID), and this variability may be simply related to small cohort size alone. To overcome this potential problem, we use a bivariate isotonic regression to smooth the resulting toxicity surface to a monotonically increasing one. The determination of the MTD contour is accomplished using the Dykstra-Roberston algorithm. Once a monotonically increasing toxicity surface is obtained (either observed or smoothed according to the bivariate isotonic regression algorithm), the MTD combinations closest to the targeted DLT rate of 0.3 but still <0.33 are calculated.

# 8.1.3. Sample Size Determination

The sample sizes planned for the study arise from logistic feasibility and past experience with Phase 1b studies in oncology and are not entirely driven by statistical considerations. It is expected that approximately 60 patients will be required to achieve all study objectives.

Due to the dynamic nature of the Bayesian allocation procedure, the sample size of the Up-and-Down design using the mTPI approach cannot be determined in advance. It is estimated 20 DLT evaluable patients will be enrolled in the dose finding stage in order to have a reliable and accurate estimate of the MTD. In addition, there will be a Dose Expansion Phase cohort to characterize safety, biomarkers, and efficacy in terms of probability (*p*) of achieving an event of interest including, but not limited to, objective response (OR). The goal will be to estimate proportions of such patients with the standard error (*SE*) of not greater than 0.08, ie, by definition,

$$SE = \sqrt{\frac{p(1-p)}{n}} \le \frac{1}{2\sqrt{n}}$$

Therefore, a sample of forty patients (n=40) in the Dose Expansion Phase cohort will allow estimation of the probability of achieving an event of interest with the standard error  $\leq 0.08$ .

The sample size estimate for the expansion cohort also takes into consideration the key tumor biomarker PD-L1 endpoints. If the observed rate of PD-L1 positives is 20% then approximately 40 patients would be required to enroll 8 PD-L1 positive patients.

# 8.2. Statistical Methods for Different Types of Endpoints

Listings and standard summary statistics will be used to analyze the study.

# **Analysis of Time-to-Event Endpoints**

Time-to-event endpoints will be summarized using the Kaplan-Meier method and displayed graphically when appropriate. Medians and two-sided 95% confidence intervals will be provided.

# **Analysis of Binary Endpoints**

Binary endpoints will be summarized by percentage rates along with the 95% confidence intervals using an exact method.

## **Analysis of Continuous Endpoints**

Continuous endpoints will be summarized by descriptive statistics, including the mean, standard deviation, median, minimum, and maximum values.

#### **Analysis of Categorical Endpoints**

The number and percentage of patients in each category will be provided for categorical variable.

## 8.3. Statistical Analyses

#### 8.3.1. Standard Analyses

- Study Conduct and Patient Disposition an accounting of the study patients in the safety analysis (SA) population will be provided. Patients not meeting the eligibility criteria will be listed. Patients not completing the study will be listed along with the reason for their discontinuation. Reasons for discontinuation will be summarized.
- **Baseline Characteristics** for patients in the SA population, characteristics such as age, height, weight, race, ethnicity, diagnosis, performance status, MSKCC risk group and medical history at study entry will be summarized in frequency tables, and descriptive statistics will be provided for quantitative variables.
- **Treatment Administration/Compliance** Administration of study medication will be presented for the SA population, by medication administered within each treatment group and will be described in terms of the duration of treatment in days (mean, median and range), number of cycles administered (mean, median and range), dose intensity,

dose modifications, dose interruptions, dose delays. Summaries for axitinib will include drug that may have been received during the lead-in PK period.

# 8.3.2. Analysis of Efficacy Endpoints

PFS, DR, and OS will be summarized using the Kaplan-Meier method and displayed graphically. The median event time and 2-sided 95% confidence interval (CI), calculated using the Brookmeyer-Crowley method, for the median will be provided for each endpoint.

Six-month and twelve-month progression-free survival (6m-PFS and 12m-PFS) will be summarized as a product limit estimator based on the Kaplan-Meier method to account for censored events, together with the corresponding 2-sided 95% CI. The 2-sided 95% CI for the log[-log(6 and 12-month PFS probabilities)] will be calculated using normal approximation and then back transformed to give the CI for the 6 and 12-month PFS rates. Analysis results will be included in the table for the PFS analysis.

The ORR will be summarized along with the corresponding exact 2-sided 95% CI calculated using a method based on the F distribution. If a patient has not achieved an objective response, but remain stable for at least 12 weeks, then the best overall response for such a patient will be SD.

For TTR, descriptive statistics including the mean (95% CI), median, and range will be provided.

Tumor Response will be presented in the form of patient data listings that include, but are not limited to, lesion type (target/non-target), received (maximum) dose, overall tumor response at each visit, and best overall response. In addition, progression date, death date, date of first response and last tumor assessment date, dates of first dose and last dose will be listed, together with DR, PFS and OS.

Listings or/and tables (when applicable) will be sorted by treatment cohort.

#### **Analysis Sets**

- Response-evaluable population for Tumor Response, PFS and OS (dose expansion cohort including the patients from the Dose Escalation Phase of the study treated at the MTD).
- Patients with an overall objective response of CR or PR in the response-evaluable population for Duration of Tumor Response and Time to Response (dose expansion cohort including the patients from the Dose Escalation Phase of the study treated at the MTD).

# 8.3.3. Analysis of Safety Endpoints

#### **Analysis Set**

Summaries and analyses of the primary safety endpoint will be based on the per
protocol analysis set. Summaries and analyses of all other safety parameters will
include all patients in the Safety Analysis Set.

- Secondary safety endpoint data will be summarized by dose level (pooling patients treated at the MTD from both phases of the study).
- Adverse events and laboratory tests will be summarized for the following study periods: entire study period and by cycle (Cycle 1, Cycle 2 and Cycles beyond 2) in the Safety Analysis Set; the PK lead-in period for those patients receiving at least one dose of axitinib during the 7 day PK lead-in period; and the treatment period starting at C1D1 for patients receiving the combination treatment.

# 8.3.3.1. Analysis of Primary Endpoint

Dose Limiting Toxicity (DLT) is the primary endpoint of the study. The occurrence of DLTs observed in the dosing cohorts is used to estimate the MTD as described in the protocol. AEs constituting DLTs will be listed per dose level.

## DLT-related listings will be produced by dose

- Patient ID.
- Dose and Date at which DLT occurred.
- Time from treatment start to onset of DLT.
- Time to resolution of DLT to Grade 1 or baseline.
- Dose interruption (yes, no).
- Time to resumption of treatment.
- DLT term.
- Action(s) taken due to DLT (stopped temporarily, permanently discontinued, no action taken, etc).

## 8.3.3.2. Analysis of Secondary Safety Endpoint

## **Adverse Events**

AEs will be graded by the Investigator according to the Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03 and coded using the Medical Dictionary for Regulatory Activities (MedDRA). The focus of AE summaries will be on treatment-emergent AEs. The number and percentage of patients who experienced any AE, serious AE (SAE), treatment-related AE, and treatment-related SAE will be summarized according to worst toxicity grades. The summaries will present AEs on the entire study period, separately for the lead-in PK period and by cycle (Cycle 1, Cycle 2 and Cycles beyond 2), as well as for the entire treatment period starting at C1D1 (first dose of MK-3475).

For AE summaries of the treatment period starting at C1D1, treatment-emergent will be defined as an adverse event with an initial onset or increasing severity after the first dose of

MK-3475. For all other AE summaries, treatment-emergent will be defined as an adverse event with an initial onset or increasing severity after the first dose of any study medication (axitinib, in the case of the lead-in PK period).

- An overall summary of AEs will be provided. The number and percentage of patients who experienced any AE, who experienced any SAE, who experienced any treatment-related AE, who experienced any treatment-related SAE, and who discontinued because of an AE will be presented. Treatment-related AEs are those judged by the investigator to be at least possibly related to the study drug (with a cause related to the study drug indicated on the CRF).
- All treatment-emergent AEs will be summarized by MedDRA SOC and preferred term. A summary of AEs by preferred term and maximum CTCAE grade will be presented. A summary of AEs by preferred term and maximum CTCAE grade group (Grade 1-2, Grade 3-4, and Grade 5) will also be presented. Treatment-emergent AEs will also be summarized for each group and pooled across the groups.
- Treatment-related AEs will be summarized by MedDRA SOC and preferred term separately for axitinib, MK-3475 and both. A summary of treatment-related AEs by preferred term and maximum CTCAE grade will be presented. A summary of treatment related AEs by preferred term and maximum CTCAE grade group (Grade 1-2 vs. Grade 3-5) will also be presented. Treatment-related AEs will also be summarized for each group and pooled across the groups.
- Deaths will be summarized by three time periods (on-treatment vs. within 90 days of end of treatment vs. > 90 days after end of treatment) and cause of death. Deaths that occurred within 28 days after the last dose of study treatment are defined as ontreatment deaths. Death data will also be listed.
- Patients who withdraw from study treatment because of an AE will be listed separately for axitinib and MK-3475. Patient discontinuation will be determined from the end of treatment (EOT) evaluation (where reason for termination is "Adverse Event") and the specific AE(s) will be determined from the AE CRF page (where action taken is "Withdrawn from Treatment").
- SAEs and treatment-related SAEs will be summarized by MedDRA SOC and preferred term. Patients who experienced a SAE will be listed.

The following analyses will be performed for AEs of special interest (including, but not limited to, hepatic disorders [ALT, AST and bilirubin], thyroid dysfunction [hypo-/hyperthyroidism], diarrhea, colitis and pneumonitis).

• Hy's Law eDISH scatterplot of Maximum ALT vs. Maximum Total Bilirubin on treatment.

- Hy's Law eDISH scatterplot of Maximum AST vs. Maximum Total Bilirubin on treatment.
- The prevalence of AEs of special interest will be summarized by preferred term and maximum CTC severity grade.
- Descriptive statistics will be presented for time to AE onset (days), time to grade 2 and grade 3/4 AE onset.

For all safety analyses, only descriptive methods will be used without any formal statistical test.

# **Laboratory Tests**

The number and percentage of patients who experienced laboratory test abnormalities will be summarized according to worst toxicity grade observed for each lab assay. The analyses will summarize laboratory tests on the entire treatment period, separately for the lead-in PK period and by cycle (Cycle 1, Cycle 2 and Cycles beyond 2), as well as for the entire treatment period starting at C1D1 (first dose of MK-3475) for patients receiving combination therapy.

For laboratory tests without CTC grade definitions, results will be categorized as normal, abnormal or not done.

- **Hematology** Descriptive statistics will be provided for each test result and for change from baseline by visit. Hematology results will be graded according to the NCI CTCAE Version 4.03. A summary of maximum CTCAE grade as well as shift summary of baseline grade by maximum CTCAE grade, cycle, and dose will be presented. Patients who developed a grade 3 or greater toxicity will also be listed.
- **Biochemistry** Descriptive statistics will be provided for each parameter result and for change from baseline by visit. Biochemistry results will be graded according to the NCI CTCAE version 4.03. A summary of maximum CTCAE grade as well as shift summary of baseline grade by maximum CTCAE grade, cycle, and dose will be presented. Patients who developed a grade 3 or greater toxicity will also be listed.
- Urine Descriptive statistics will be provided for urine protein and blood results and for change from baseline by visit. Urine protein and blood data will also be listed and patients with urine protein ≥2+ by semiquantitative method (e.g., dipstick) will have their 24 hour urine collection protein levels listed as well. A shift summary of baseline value by maximum value, cycle and dose will be presented for urine protein.
- Other Laboratory Tests Individual patient test results will be listed.

## **ECOG Performance Status**

ECOG performance status data will be summarized with a shift table of the baseline and the worst on study status. Baseline will be defined as the last evaluation within 28 days prior to the first dose of either axitinib or MK-3475, whichever occurs first.

# Vital Signs

Summaries and listings will be presented for blood pressure, body weight and pulse rate.

In addition, the baseline and the change from baseline in blood pressure and pulse rate will be summarized using descriptive statistics by visit. Baseline will be defined as the last evaluation within 28 days prior to the first dose of either axitinib or MK-3475, whichever occurs first.

## **ECG**

All ECG measurements obtained during the study will be listed. Single ECG measurements will be obtained at screening and on Cycle 1 Day 1 and End of Treatment/Withdrawal as well as when clinically indicated.

# **Concomitant Medications and Non-drug Procedure/Treatments**

All drug medications will be coded by the World Health Organization (WHO) medical dictionary. Non-drug procedure/treatments will be coded by the MedDRA dictionary. All medications with a start date prior to lead-in D1 (for patients with a lead-in period) or prior to C1D1 (for patients with no lead-in period) are considered previous medication. All ongoing medications at the end of study or medications with a stop date on or after lead-in D1 (for patients with a lead-in period) or prior to C1D1 (for patients with no lead-in period) are considered concomitant medication. If a medication satisfies both the definition of previous and concomitant medication, it will be considered both previous and concomitant medication

The number of subjects with any concomitant drug/non-drug treatment will be summarized. Listings of prior and concomitant drug/non-drug treatment will be provided separately. If any prior or concurrent surgery or radiation therapy is given, these data will be listed for each patient. Furthermore, follow-up systemic therapy for the primary diagnosis will be summarized by categories of follow-up therapy and will be listed for each patient as appropriate.

#### **Data Safety Monitoring Committee**

A Data Safety Monitoring Committee will not be established for the study.

## 8.3.4. Analysis of Pharmacokinetics

Analysis Set: PK

#### 8.3.4.1. Pharmacokinetic Analysis of MK-3475 and Axitinib

Standard PK parameters for axitinib ( $C_{max}$ ,  $T_{max}$ ,  $AUC_{0-last}$ ,  $AUC_{0-12}$ ,  $AUC_{0-24}$ , CL/F, Vz/F, and plasma elimination half life  $t_{1/2}$ ) will be estimated using non-compartmental methods. For MK-3475, pharmacokinetics will be evaluated at Merck using population pharmacokinetic modeling and results will be shared with pfizer.

Presentation of pharmacokinetic data will include:

- Descriptive statistics (n, mean, SD, %CV, median, minimum, maximum) of plasma concentrations for axitinib will be presented in tabular form by treatment cohort, dose level, cycle, day and nominal time. Additionally similar descriptive statistics will also be generated for dose-normalized axitinib pharmacokinetic parameters
- Linear-linear and log-linear plots of mean and median plasma concentrations by nominal time for axitinib will be presented for PK sampling days by treatment cohort, cycle, and study day. Similar plots will be presented for axitinib for each individual patient concentrations. Only patients who have matched pairs of PK collections available on both planned treatments (when administered alone and in combination with MK-3475) will be included in the axitinib plasma concentration descriptive summary and median concentration profiles. Patients who have undergone intrapatient dose reduction or escalation will be excluded from the median plasma concentration-time plots.
- Pharmacokinetic parameters for axitinib will be listed and summarized by treatment cohort/dose level, cycle and study day using descriptive statistics (n, mean, SD, %CV, median, minimum, maximum, geometric mean and its associated %CV, and 95% confidence interval). For Tmax, the range (min, max) will be also be provided. Only patients who have a matched pair of estimated axitinib PK parameters available on both planned treatments (when administered alone and in combination) will be included in the axitinib PK parameter summary tables. PK parameters with zero values will be excluded from the calculation of geometric means and its associated %CV. If an intra patient dose escalation or reduction occurs, dose-dependent PK parameters (AUC and C<sub>max</sub>) for that patient may be dose-normalized when it is known that the drug exhibits linear PK within the dose range and other PK parameters will be reported as estimated; or may only be included in descriptive statistics and summary plots up to the time of the dose change. In addition, dose-normalized axitinib C<sub>max</sub> and AUC parameters will be summarized (as described above) using data pooled across cohorts in which different axitinib doses were administered.
- Box plots for AUC and C<sub>max</sub> for axitinib (during treatments when given alone and in combination) will be generated. Individual data points, the geometric mean and the median of the parameter in each treatment will be overlaid on the box plots. If a cohort has limited evaluable PK data (n<4), matchstick plots showing changes in AUC and C<sub>max</sub> for each drug (during treatments when given alone and in combination) in individual patients will then be generated. The geometric mean of the parameter in each treatment will be overlaid in the plots. In addition, box plots

for dose-normalized axitinib  $C_{max}$  and AUC parameters will be created using data pooled across cohorts in which different axitinib doses were administered.

 Trough concentrations for MK-3475, if available, will be plotted for each treatment cohort using a box-whisker plot by cycle and day within cycle in order to assess the attainment of steady-state.

#### 8.3.4.2. Effect of MK-3475 on Axitinib Pharmacokinetics

The effect of repeated MK-3475 dosing on steady-state axitinib PK will be evaluated using  $AUC_{0-12}$  (or  $AUC_{0-last}$ , if  $AUC_{0-12}$  is not estimable) of axitinib on Lead-in Day 7 and Cycle 7 Day 1, respectively, as the primary PK parameter. Ninety-percent confidence interval for the ratio of geometric means of  $AUC_{0-12}$  and Cmax (axitinib in presence of MK-3475/axitinib alone) will be computed to assess the magnitude of the effect.

## 8.3.4.3. Immunogenecity Assessment

Results for the anti-MK-3475 antibody (ADA) assessment will be provided by Merck.

# 8.3.4.4. Population Pharmacokinetic Analysis or PK/PD Modeling

Mechanism-based or semi-mechanistic sequential pharmacokinetic-pharmacodynamic models may be developed using NONMEM® to explore any relationships between plasma drug concentrations and selected safety, biomarker, and efficacy endpoints.

The results of these analyses, if performed, will be reported separately.

# 8.3.5. Analysis of Biomarker Endpoints

Translational and pharmacodynamic biomarkers will be summarized using the appropriate biomarker analysis set. Summaries of baseline and ratio to baseline values at post-treatment visits will be provided using N, mean, standard deviation, median, % CV (as appropriate) and minimum/maximum for circulating biomarkers serum and tumor RNA measurements for potential gene signature development. Summary statistics will be provided for baseline values of circulating markers including VEGF-A, VEGFR2, IL8 and T-cell receptors, and archival tumor and baseline *de novo* biospecimens markers such as PD-L1 for all biomarker evaluable patients. Post-baseline values will be summarized for biomarker evaluable patients in the dose expansion cohort, when available.

Correlations of biomarker results with measures of anti-tumor efficacy will be examined for dose escalation and expansion cohorts separately. Summary of level of biomarkers at baseline and/or ratio of values to baseline versus ORR category will be made by timepoint. Summary of PFS and DR will be provided for dose expansion cohort after stratification by a preset cutpoint of biomarker values at baseline and/or ratio of values to baseline by timepoint. Receiver Operating Characteristics (ROC) analysis may be conducted for significant test results (p<0.05) in correlations of PFS and/or ORR with PD-L1 expression level. Receiver Operating Characteristics (ROC) analysis may also be performed if significant test results (p<0.05) in correlations of ORR and/or PFS with tumor RNA measurements are observed.

Graphical display will be provided for level of biomarkers at baseline and/or ratio of values

to baseline at each timepoint. Box and Whisker plots will be produced for level of biomarkers at baseline and/or ratio of values to baseline versus ORR category by timepoint in dose escalation and expansion cohorts separately. Kaplan-Meier plots will be produced for PFS and DR after stratification by < or >= median levels of biomarkers at baseline and/or ratio of values to baseline at each timepoint in the dose expansion cohort.

All biomarker data will be listed.

# 8.4. Summary of Secondary Efficacy Analyses

| Endpoint | Analysis<br>Population | Statistical Method | Missing Data | Analysis<br>Type/Timing |
|---|---|---|---|---|
| ORR | Response<br>Evaluable | Exact method based on F-distribution (95% CI) (See 8.3.2) | See Section 6.1 | Secondary<br>analysis |
| DR | Subgroup of<br>pts with OR<br>from the<br>Response<br>Evaluable | K-M method (median and 95% CI) (See 8.3.2) | See Section 6.1 | Secondary<br>analysis |
| TTR | Response<br>Evaluable | Univariate (median and 95% CI) (See 8.3.2) | See Section 6.1 | Secondary<br>analysis |
| PFS | Response<br>Evaluable | K-M method (median, 6 and 12m-PFS and 95% CIs) (See 8.3.2) | Censor patients on<br>the day of the last<br>evaluable tumor<br>assessment<br>documenting<br>absence of disease<br>progression for<br>(See Section 6.1) | Secondary<br>analysis |
| OS Response<br>Evaluable | | K-M method (median<br>and 95% CIs)<br>(See 8.3.2) | See Section 6.1 | Secondary<br>analysis |

CI: Confidence intervals; DR: Duration of Response; K-M: Kaplan-Meier; OR: Objective Response; ORR: Objective Response Rate; PFS: Progression-free Survival; TTR: Time to Response; OS: Overall Survival

## 9. REFERENCES

- 1. Brookmeyer R, Crowley JJ. A confidence interval for the median survival time. Biometrics. 38: 29-41, 1982.
- 2. Kaplan EL, Meier P. Nonparametric estimation from incomplete observations. J Am Stat Assoc. 53: 457-81, 1958.
- 3. Eisenhauer EA, Therasse P, Bogaerts J, et al. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47.
- 4. Fanale M et al. Phase I study of bortezomib plus ICE (BICE) for the treatment of relapsed/refractory Hodgkin lymphoma. British Journal of Haematology, 154:284 286, 2011.
- 5. Ji Y et al. A modified toxicity probability interval method for dose-finding trials. Clinical Trials 2010; 7:653 663.
- 6. Dykstra R, Robertson T. An algorithm for isotonic regression for two or more independent variables. *Ann Stat.* 1982;10:708-716.

#### 10. APPENDICES

# Appendix 1. Programming Specifications for AE Analyses

#### a. Time to AE onset

#### 1. Definition

Time to AE onset (days) will be calculated as first AE start date – first dose date +1. The definition and calculations are similar for time to Grade 3/4 AE onset.

#### AE start date

The Date of Onset for the first occurrence of the AE based on the Log AE CRF page.

#### *First dose date*

For AE summaries of the lead-in PK period: The date of the first dose taken from the Axitinib Dosing CRF page.

For AE summaries of the treatment period starting at C1D1: The date of the first dose taken from the MK-3475 Dosing CRF page.

For AE summaries of the entire treatment period (including by cycle): The date of the first dose taken from either the Axitinib or MK-3475 Dosing CRF page, whichever occurs first.

## b. Duration of AE

#### 1. Definition

Duration of AE (days) is defined as the cumulative duration across episodes of the specific AE (by preferred terms) where duration for each episode is calculated as AE end date – AE start date +1 excluding any overlap. Duration of AE is defined for subjects with the AE.

#### AE start date

The Date of Onset based on the Log AE CRF page.

## AE end date

The Date Resolved based on the Log AE CRF page.

#### 2. Censoring

AE resolution is considered an event (censoring variable=1). If a subject has an AE that was ongoing (does not have to be the last AE) at the time of analysis, the time is censored (censoring variable=0) at the last available on treatment visit date. Subjects who die prior to resolution of the AE will be censored at the *date of death*. If the date of death is the same as the date of the resolution of the AE, the subject will be censored at that date (i.e. resolution will not be considered an event) and only if the AE is the AE that resulted in death will it be counted as an event.

#### Date of death

Death date is based on the Notice of Death CRF page.

#### 3. Clustered Events

For clustered events, a patient could have multiple events in the cluster which may overlap. In this case, AE duration will be summed across all events in the cluster accounting for the overlap (i.e. overlapping periods between events in the same cluster are not double-counted). Lags between events in the same cluster are not included in the duration.

The following scenarios provide examples of the calculation for 2 events in the same cluster. The extension to 3 or more events of the same cluster is similar.

# • TWO EVENTS OF THE SAME CLUSTER WHERE ONE EVENT COMPLETELY CONTAINS THE OTHER EVENT

| event 1 | [ | ] |
|---------------|----------------------|----------|
| | startda | enddate1 |
| event 2 | [ | ] |
| | startdate2 | enddate2 |
| duration = en | nddate1-startdate1+1 | |

#### CERTAIN PORTIONS OF TWO EVENTS IN THE SAME CLUSTER OVERLAP



duration = enddate2-startdate1+1

## • TWO EVENTS OF THE SAME CLUSTER ARE CONTIGUOUS TO EACH OTHER



duration = enddate2-startdate1+1

| • | TWA EVENTS | OF THE CAME | CHUCTED | ARE NON-OVERI | A DDING |
|---|------------|-------------|---------|---------------|---------|
| • | | OF THE SAME | CLUSIER | ARE NUN-UVERI | AFFHNU |

| event I | L | ] | | |
|---|---|---|---|---|
| | startdate1 | enddate1 | | |
| event 2 | | | [ | ] |
| | | | startdate2 | enddate2 |
| duration = (endda | te1-startdate1+1) + (e | nddate2-starta | late2+1) | |

# c. AE Prevalence

#### 1. Definition

AE prevalence is defined as the number of patients with an AE in a particular time period (including both new cases with an onset date during the specified time period AND cases with an AE continued from a previous time period) divided by the number of patients at risk during the specified time period. The number of patients at risk includes all subjects except those who either have discontinued or died prior to the specified time period.

AE prevalence will be presented for the entire study period, separately for the lead-in PK period and by cycle (Cycle 1, Cycle 2 and Cycles beyond 2), as well as for the entire treatment period starting at C1D1.

#### 2. Assumptions

For AE summaries of the study period starting at C1D1 the following apply:

- A patient is counted in the numerator if the patient has an onset date of the AE during Cycle 1 OR for patients with a 7 day lead-in PK period there is an increase in grade of the AE after the first dose of MK-3475 (C1D1) or if there is a decrease and then subsequent increase during treatment with the combination.
- The denominator will include subjects who have received at least one dose of MK-3475.

For AE summaries of the entire study period including by cycle (Lead-in PK period, Cycle 1, Cycle 2 and Cycles beyond 2) the following apply:

- Patients are counted for an AE in each cycle up until the cycle where the AE resolved. Thus, the calculation conservatively assumes that if the AE resolved in a cycle, it resolved at the end of the cycle.
- For Lead-in PK period, a patient is counted in the numerator if the patient has an onset date of the AE during the Lead-in period.
- For Cycle 1, a patient is counted in the numerator if the patient has an onset date of the AE during Cycle 1 OR an onset date during the Lead-in PK phase that is still ongoing in Cycle 1 (did not have a resolution date in the Lead-in phase).
- For Cycle 2, a patient is counted in the numerator if the patient has an onset date of the AE during Cycle 2 OR an onset date during the Lead-in PK phase or Cycle 1 that is still ongoing in Cycle 2 (did not have a resolution date in the Lead-in phase or Cycle 1).

- For Cycles ≥2, a patient is counted in the numerator if the patient has an onset date in Cycles ≥2 OR an onset date in a previous cycle that is still ongoing (did not have a resolution date in Cycle 1 or earlier).
- The denominator for a particular time period will include subjects who are at risk prior to the time period. The number at risk includes all subjects except those who either have discontinued (based on the 'Subject Summary' CRF) or died prior to the specified time period (i.e. Death Date based on 'Notice of Death' CRF is prior to start of time period).

# **Appendix 2. Study Specific Information for Efficacy**

• **Baseline**: is defined as the last observation within 28 days prior to the first dose of any study treatment (first dose of axitinib for patients receiving the lead-in PK dose or first dose of either drug for patients not receiving the lead-in PK dose).

# • Adequate Baseline:

- Baseline tumor evaluations must be performed within 4 weeks (28 days) prior to the first dose of any study treatment (first dose of axitinib for patients receiving the lead-in PK dose or first dose of either drug for patients not receiving the leadin PK dose);
- Presence of at least one measurable lesion per RECIST version 1.1;
- All lesions recorded at baseline must have an associated status recorded on the CRF;
- Baseline lesions must be assessed with an acceptable method that includes:
   Conventional CT Scan, Spiral CT Scan, X-ray, MRI, Physical Exam, Bone Scan
   and Other. Note: If based on data review "unacceptable" methods (e.g.
   ultrasound, etc) are noted under "Other", then this category will not be considered
   acceptable (on a case by case basis).
- "On-study" period for efficacy: is defined as the period from the date of the first dose of MK-3475 until subject death, progression of disease, subject no longer willing to participate, start of other anti-cancer treatment,, whichever is earlier.
- **Subsequent anti-tumor treatment:** includes any systemic anticancer therapy (other than study medication), radiation to target lesions, and surgery for removal (resected or partially resected) of target lesions.

# Appendix 3. RECIST 1.1

The determination of antitumor efficacy during this study will be based on objective tumor assessments made according to the RECIST system of unidimensional evaluation.

# **Measurability of Tumor Lesions**

At baseline, individual tumor lesions will be categorized by the Investigator as either measurable or non-measurable by the RECIST criteria as described below.

#### Measurable:

<u>Tumor lesion</u>: Must be accurately measured in at least one dimension (longest diameter in the plane of measurement is to be recorded) with a minimum size of:

- 10 mm by CT scan (CT scan slice thickness no greater than 5 mm);
- 10 mm caliper measurement by clinical exam (lesions which cannot be accurately measured with calipers should be recorded as non-measurable).

Malignant lymph nodes: To be considered pathologically enlarged and measurable, a lymph node must be ≥15mm in short axis when assessed by CT scan (CT scan slice thickness recommended to be no greater than 5 mm). At baseline and in follow-up, only the short axis will be measured and followed.

**Non-Measurable:** All other lesions, including small lesions (longest diameter <10mm or pathological lymph nodes with  $\ge 10$  mm to <15 mm short axis) as well as truly non-measurable lesions. Lesions considered truly non-measurable include: leptomeningeal disease, ascites, pleural or pericardial effusion, inflammatory breast disease, lymphangitic involvement of skin or lung, abdominal masses/abdominal organomegaly identified by physical exam that is not measurable by reproducible imaging techniques.

NOTE: If measurable disease is restricted to a solitary lesion, its neoplastic nature should be confirmed by cytology/histology.

# **Recording Tumor Measurements**

All measurable lesions up to a maximum of 2 lesions per organ and 5 lesions in total representative of all involved organs should be identified as **target lesions** and measured and recorded at baseline and at the stipulated intervals during treatment. Target lesions should be selected on the basis of their size (lesion with the longest diameters) and their suitability for accurate repetitive measurements (either by imaging techniques or clinically).

The longest diameter will be recorded for each target lesion. The sum of the longest diameter for all target lesions will be calculated and recorded as the baseline sum longest diameter to be used as reference to further characterize the objective tumor response of the measurable dimension of the disease during treatment. All measurements should be performed using a caliper or ruler and should be recorded in metric notation in centimeters.

All other lesions (or sites of disease) should be identified as **non-target lesions** and should also be recorded at baseline. Measurements are not required and these lesions should be followed as "present" or "absent."

# **Techniques for Assessing Measurable Disease**

The same method of assessment and the same technique should be used to characterize each identified and reported lesion at screening and during follow-up. Imaging-based evaluation is preferred to evaluation by clinical (physical) examination when both methods have been used to assess the antitumor effect of a treatment.

# **Definitions of Tumor Response**

# **Target Lesions**

**Complete response (CR)** is defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm

**Partial response (PR)** is defined as a  $\geq 30\%$  decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions.

**Progressive disease (PD)** is defined as a  $\geq 20\%$  increase in the sum of the longest dimensions of the target lesions taking as a reference the smallest sum of the longest dimensions recorded since the treatment started, or the appearance of one or more new lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.

**Stable disease (SD)** is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as a reference the smallest sum of the longest dimensions since the treatment started.

# **Non-Target Lesions**

Complete response (CR) is defined as the disappearance of all non-target lesions. All lymph nodes must be non-pathological in size (<10mm short axis).

**Non-CR/Non-PD** is defined as a persistence of  $\geq 1$  non-target lesions.

**Progressive disease (PD)** is defined as unequivocal progression of existing non-target lesions, or the appearance of  $\geq 1$  new lesion.

The cytological confirmation of the neoplastic origin of any effusion that appears or worsens during treatment when the measurable tumor has met criteria for response or stable disease is mandatory to differentiate between response or stable disease and progressive disease.

# **Confirmation of Tumor Response**

To be assigned a status of PR or CR, changes in tumor measurements in patients with responding tumors must be confirmed by repeat studies that should be performed ≥4 weeks after the criteria for response are first met. In the case of SD, follow-up measurements must have met the SD criteria at least once after study entry at a minimum interval of 12 weeks.

#### **Determination of Tumor Response by the RECIST Criteria**

When both target and non-target lesions are present, individual assessments will be recorded separately. Determination of tumor response at each assessment is summarized in the following table.

# Response Evaluation Criteria in Solid Tumors

| Target Lesions <sup>1</sup> | Non-Target Lesions <sup>2</sup> | New Lesions <sup>3</sup> | Tumor Response |
|---|---|---|---|
| CR | CR | No | CR |
| CR | Non-CR/non-PD | No | PR |
| CR | Not evaluated | No | PR |
| PR | Non-PD or not all evaluated | No | PR |
| SD | Non-PD or not all evaluated | No | SD |
| PD | Any response | Yes or No | PD |
| Any response | PD | Yes or No | PD |
| Any response | Any response | Yes | PD |

<sup>1</sup> Measurable lesions only.

# **Determination of Best Overall Response**

The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started). For CR and PR, the patient's best response assignment will depend on the achievement of both measurement and confirmation criteria. In the case of SD, follow-up measurements must have met the SD criteria at least once after study entry at a minimum interval of 12 weeks.

NOTE: Patients with a global deterioration of health status requiring discontinuation of treatment without objective evidence of disease progression at that time should be reported as "symptomatic deterioration." Every effort should be made to document the objective progression even after discontinuation of treatment. It should also be noted that a tumor marker increase does not constitute adequate objective evidence of tumor progression. However, such a tumor marker increase should prompt a repeat radiographic evaluation to document whether or not objective tumor progression has occurred.

In some circumstances, it may be difficult to distinguish residual disease from normal tissue. When the evaluation of complete response depends upon this determination, it is recommended that the residual lesion be investigated by fine needle aspirate or biopsy before confirming the complete response status.

<sup>&</sup>lt;sup>2</sup> May include measurable lesions not followed as target lesions or non-measurable lesions.

<sup>&</sup>lt;sup>3</sup> Measurable or non-measurable lesions

Appendix 4. Detailed Dose Escalation/De-Escalation Scheme

| | | Number of patients treated at current dose | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| | 0 | E | E | E | E | E | E | E | E | E | E |
| | 1 | D | $\mathbf{S}$ | S | $\mathbf{S}$ | $\mathbf{S}$ | E | E | E | E | E |
| ø | 2 | | $\mathbf{D}\mathbf{U}$ | D | S | S | $\mathbf{S}$ | S | S | $\mathbf{S}$ | S |
| Number of toxicities | 3 | | | $\mathbf{D}\mathbf{U}$ | DU | D | D | $\mathbf{S}$ | $\mathbf{S}$ | $\mathbf{S}$ | S |
| toxi | 4 | | | | $\mathbf{D}\mathbf{U}$ | DU | DU | DU | DU | DU | DU |
| . of 1 | 5 | | | | | DU | DU | DU | DU | DU | DU |
| ıber | 6 | | | | | | $\mathbf{DU}$ | DU | DU | DU | DU |
| _ un | 7 | | | | | | | DU | DU | DU | DU |
| | 8 | | | | | | | | DU | DU | DU |
| | 9 | | | | | | | | | DU | DU |
| | 10 | | | | | | | | | | DU |

**E** = Escalate to the next higher dose **S** = Stay at the current dose

D = De-escalate to the next lower dose

U = The current dose is unacceptably toxic

MTD = 30%